CLINICAL TRIAL: NCT02611102
Title: Effects of Daily Butter & Medium-Chain Triglyceride Oil on Lipoproteins When Added to Baseline Diet a Randomized Controlled Trial
Brief Title: Effect of Butter & MCT Oil on Lipoproteins - A RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 404482-2
Record Dates: First submitted 2015-06-10; First posted 2015-11-20 (Estimated); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Hyperlipidemia
Keywords: cardiovascular disease/medium-chain-triglycerides/cholesterol
MeSH Terms: conditions — Hyperlipidemias; Cardiovascular Diseases | interventions — Butter; Coffee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MCT oil + Butter in Coffee (Experimental): This group will be provided with MCT oil and butter to add to their daily coffee intake.
  Interventions: Dietary Supplement: MCT oil + Butter in Coffee
- Low calorie coffee (Placebo Comparator): This group will continue to drink their normal daily coffee with < 50kcal of creamer and/or sweetener.
  Interventions: Dietary Supplement: MCT oil + Butter in Coffee

INTERVENTIONS:
Dietary Supplement: MCT oil + Butter in Coffee — 2 tablespoons medium-chain triglyceride oil + 2 tablespoons butter added to 2-4 cups of coffee similar to their usual intake prior to 1200 daily over a 4 week period after a 2 week run-in phase during which the doses of butter and MCT oil will be titrated up (1 Tbsp. of each butter + MCT x 5 days, 2 Tbsp. butter + 1 Tbsp. MCT x 5 days, then 2 Tbsp. of each x 4 days) followed by 6 weeks of washout without treatment.

SUMMARY:
Determine the effects on lipoprotein profiles of high dose concentrated dietary SFA (saturated fatty acids) (from MCT (medium-chain triglyceride) oil + butter) in combination added to coffee. The study will be conducted as a RCT in healthy adults without cardiometabolic disease or conditions that influence lipoprotein metabolism or other specific dietary recommendations.

DETAILED DESCRIPTION:
Research Design A prospective randomized controlled interventional study

Methodology /Technical Approach A total of up to 60 subjects will be recruited to allow for completion of the study by a minimum of 17 subjects per arm. Subjects will be randomized to one of two groups in a 1:1 ratio. Recruited subjects will be adult coffee drinkers between the ages of 18-45 without hyperlipidemia and without criteria for diabetes or pre-diabetes. Subjects will have baseline weight, waist circumference (WC), and blood-pressure (BP) measurements obtained. Subjects will have baseline fasting lipids,, CMP,HbA1c,TSH,and hsCRP. The subjects will be stratified by gender and randomized to receive one of two dietary regimens: 1) coffee (< 50 kcal of added creamer/sweetener) or 2) coffee with butter + medium-chain triglyceride (MCT) oil combination (2 tbsp. MCT containing 230kcal and 28gm fat+ 2 tbsp butter containing 200kcal and 22gm fat). The drink will be consumed daily over a 4 week period. Dietary history will be evaluated by via the ASA24website (http://appliedresearch.cancer.gov/asa24/). At 6 and 12 weeks post-consent, baseline labs will be repeated. The primary outcome is change in apolipoprotein B between groups. Secondary outcomes include changes in lipids, WC, BP, HbA1c, and FBG. Exploratory analysis will include changes in dietary macronutrient load and subgroup analysis of effects related to dietary patterns.

Primary objective:

1. Evaluate clinically and statistically significant changes of apoB number in healthy adults who consume coffee with butter and MCT oil.

Secondary objectives:

1. Evaluating change in:

1. non-HDL-c
2. LDL-c
3. triglycerides
4. BP
5. waist circumference
6. FBG
7. HbA1c

Exploratory objective:

1. Change in macronutrient profiles of dietary patterns.

Our null hypothesis is that the addition of butter and medium-chain triglyceride oil at proposed doses has no clinically significant effects on atherogenic lipoproteins, namely apo lipoprotein B particles (apoB).

ELIGIBILITY:
Inclusion Criteria:

1. DoD healthcare beneficiaries
2. willing to drink 2 to 4 cups of coffee daily
3. between the ages of 18 to 45
4. serum LDL-c < 160,
5. non-HDL-c < 190
6. apoB < 120

Exclusion Criteria:

1. BMI > 30kg/m2 or < 20kg/m2 or waist circumference > 102cm (males) or 88cm (females)
2. Triglycerides > 150
3. Hypertension defined as SBP > 150, DBP > 90 or on treatment for high blood pressure
4. Chronic liver disease defined by any clinical or a history of serum AST or ALT > 3 times ULN
5. Kidney disease defined as a GFR <90 ml/min or history of nephritic syndrome
6. Impaired glucose metabolism defined as HbA1c > 5.6, FBG > 99, or 2-hour OGTT > 139
7. Any known malignancy
8. Known malabsorption disorder to include inflammatory bowel disease, celiac disease, cystic fibrosis, history of gastric bypass
9. Hypothyroidism per lab evaluation at baseline
10. Pregnancy
11. Polycystic Ovary Syndrome or irregular menstrual periods
12. Subjects taking certain medications such as glucocorticoids, immunosuppressants (cyclosporine, sirolimus, etc.), tamoxifen, androgens, antipsychotics, hydrochlorothiazide, retinoids, beta-blockers, statins, bile acid sequestrants, niacin, fibrates, ezetimibe, high dose fish oil (>1gm/day epa + dha), or any other supplement or pharmacologic agent known to alter lipoproteins

    a. If on hormonal contraceptives, lipid panel must be stable over the past 12-24 months
13. Cushing's syndrome per medical history or clinical suspicion
14. HIV per medical history
15. Chronic Inflammatory Disorders such as, but not limited to, SLE, RA, IBD per medical history
16. History of tobacco use within the previous 12 months to include cigarettes, e-cigarettes, chewing tobacco, cigars, and pipes.
17. History of marijuana use within the previous 12 months
18. Active intentional weight loss of over 5% in the past 3 months

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2016-03-08 (Actual); Primary Completion 2022-03 (Actual); Study Completion 2022-03 (Actual)

PRIMARY OUTCOMES:
Changes in apolipoprotein B | Baseline and 6 weeks
  Evaluate clinically and statistically significant changes of apoB number in healthy adults who consume coffee with butter and MCT oil.

SECONDARY OUTCOMES:
non-HDL-c | 6 weeks
  Evaluating change in non-HDL_c
LDL-c | 6 weeks
  Evaluating change in LDL-c
triglycerides | 6 weeks
  Evaluating change in triglycerides
Blood pressure | 6 weeks
  Evaluating change in blood pressure
waist circumference | 6 weeks
  Evaluating change in waist circumference
Fasting Blood Glucose | 6 weeks
  Evaluating change in fasting blood glucose
HbA1c | 6 weeks
  Evaluating change in HbA1c

CONTACTS AND LOCATIONS:
Overall Officials: Thanh D Hoang, DO, Principal Investigator — WRNMMC
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States